CLINICAL TRIAL: NCT04296019
Title: A Randomized, Open-label, Multicenter, Phase II Clinical Study Evaluating the Efficacy and Safety of Fruquintinib as a Maintenance Therapy Following First-line Treatment for Metastatic Colorectal Cancer
Brief Title: Fruquintinib as a Maintenance Therapy Following First-line Treatment for Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-ON-09
Record Dates: First submitted 2020-01-01; First posted 2020-03-05 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Colo-rectal Cancer
Keywords: fruquintinib; Colo-rectal Cancer; maintenance therapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fruquintinib (Experimental): Patients who achieved stable disease (SD) or partial response (PR) or complete response (CR) following palliative first-line treatment will receive maintenance therapy with fruquintinib.
  Interventions: Drug: Fruquintinib
- Observation (No Intervention): Patients who achieved SD or PR or CR following palliative first-line treatment will receive treatment-free observation.

INTERVENTIONS:
Drug: Fruquintinib — Maintenance therapy with fruquintinib ( 5 mg qd for 3 consecutive weeks, followed by discontinuation for 1 week).
  Arms: Fruquintinib

SUMMARY:
This study was a randomized, controled, multicenter, phase II clinical study evaluating the efficacy and safety of fruquintinib as a maintenance therapy following first-line treatment for metastatic colorectal cancer. This study will include the patients with confirmed unresectable metastatic left-sided colon cancer with RAS mutation or right-sided colon cancer who achieved stable disease (SD) or partial response (PR) or complete response (CR) via palliative first-line treatment. It's expected to include 110 patients and they will be randomly stratified at 2:1 into fruquintinib group and observation group based on whether bevacizumab is used and the primary tumor site, using the Interactive Network Response System (IWRS). The random No. corresponds to the respective patient. The enrollment time is expected to be 18 months, followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old (including 18 and 75 years);
* Eastern Cooperative Oncology Group-performance score (ECOG PS) 0 or 1;
* Estimated survival ≥ 6 months;
* Histologically and/or cytologically confirmed metastatic left-sided colon cancer with RAS mutation or right-sided colon cancer, having unresectable metastatic or recurrent foci;
* Having received first-line systemic anti-tumor therapy for mCRC (chemotherapeutic drugs may include fluorouracil, oxaliplatin, irinotecan, such as XELOX, FOLFOX, FOLFIRI, and can combine or not combine with bevacizumab); achieving RECIST1.1-assessed SD (stable disease) or PR (partial response) or CR (complete response) after 18-24 weeks of first-line treatment.
* UCG suggesting left ventricular ejection fraction ≥50%;
* Having fully understood and voluntarily signed the informed consent.

Exclusion Criteria:

* Absolute neutrophil count (ANC) <1.5×109/L, or platelet count <80×109/L, or hemoglobin < 9g/dL; it's not allowed to perform blood transfusion within 2 week before enrollment to meet the inclusion criteria;
* Serum total bilirubin > 1.5 × upper limit of normal (ULN); > 2.5 × ULN for patients with hepatic metastases;
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) > 2.5 × ULN, or > 5 × ULN for patients with hepatic metastases;
* Serum creatinine > 1.5 × upper limit of normal (ULN), or creatinine clearance < 50mL / min (calculated using Cockcroft-Gault formula);
* Partial prothrombin time (APTT) or prothrombin time (PT) > 1.5 times ULN (based on the normal value in the clinical study center);
* Clinically significant electrolyte abnormalities;
* Urine protein 2+ or above, or 24-hour urinary protein quantity ≥ 1.0g / 24h;
* Subjects with dysphagia or known drug absorption disorders;
* Presence of brain metastasis or leptomeningeal metastasis;
* The toxicity of previous anticancer treatment has not yet reduced to (NCI CTC AE) level 1, excluding alopecia and oxaliplatin-induced neurotoxicity ≤ 2); patients haven't not fully recovered from previous surgery or less than 4 weeks elapsed since previous anticancer treatment or surgery;
* Patients have clinically detectable second primary malignant tumors at enrollment, or have other malignant tumors (except for well-treated basal cell carcinoma or cervical carcinoma in situ) in the past 5 years;
* Patients have clinically uncontrolled active infections such as acute pneumonia, hepatitis B or hepatitis C activity (previous history of hepatitis B infection, whether or not under medication control, HBV DNA ≥ 104 copies or ≥ 2000 IU/ml);
* Patients have hypertension that cannot be controlled by a single drug. That is, after single drug treatment, systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg;
* Patients currently have digestive tract diseases such as duodenal ulcer, ulcerative colitis, intestinal obstruction or other conditions that may cause gastrointestinal bleeding or perforation at the discretion of the investigator; or patients have undergone surgery for intestinal perforation and intestinal fistula but was uncured.
* Patients have a history of arterial thrombosis or deep vein thrombosis within 6 months prior to enrollment, or patients have bleeding tendency or bleeding history within the 2 months before enrollment, regardless of severity;
* Patients have a stroke or transient ischemic attack within 12 months prior to enrollment;
* Skin wounds, surgical sites, trauma site, severe mucosal ulcers or fractures haven't completely healed yet.
* Patients have acute myocardial infarction, severe/unstable angina, coronary artery bypass grafting or NYHA Class II/more severe cardiac insufficiency within 6 months prior to enrollment;
* Pregnant or lactating women; or women with potentiality of childbearing have a positive pregnancy test result before the first dose;
* Patients have any clinical or laboratory abnormalities or compliance problems so that the investigator believes that they are not suitable to participate in this clinical study;
* Patients have serious psychological or mental abnormalities;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
PFS | 24 months after the last subject participating in
  progression-free survival (PFS) is defined as time from randomization to disease progression.

SECONDARY OUTCOMES:
OS | 36 months after the last subject participating in
  Overall survival (OS) is defined as time from randomization to death.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 month after the last administration of fruquintinib
  Adverse events (AE) will be graded and documented according to NCI-CTC AE v4.0 from the beginning of treatment to 1 months after the last date of treatment. Documentary will include severity, lasting period and occurrence time. Main AEs include hypertension, albuminuria, skin reaction of hands and feet, hemorrhage, dysphonia, transaminase rise, abdominal pain / abdominal discomfort, blood bilirubin rise, thyroid dysfunction, infection, diarrhea, fatigue / fatigue, appetite decline, oral mucositis, weight loss, fecal occult blood and platelet count decline

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China